CLINICAL TRIAL: NCT01194544
Title: The Relationship Between Dietary Habit and Gastroesophageal Flap Valve Abnormality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Yung-Fa Chen M.D., Taipei Medical University WanFang Hospital
Other Study IDs: 99033
Record Dates: First submitted 2010-08-10; First posted 2010-09-03 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- population undergoing EGD in health examination.

SUMMARY:
Gastroesophageal reflux disease (GERD) is commonly seen in Western countries; however, it is gaining prevalence in Asia countries recently. In addition to the lower esophageal sphincter and the crural fibers of the diaphragm, the flap valve at the gastroesophageal junction is also responsible for maintaining an antireflux barrier. Hill et al developed a grading system of gastroesophageal flap valve (GEFV) and concluded that this flap valve system is simple, reproducible, and offers diagnostic aid in the evaluation of patients with suspicious reflux disease undergoing esophagogastroduodenoscopy (EGD). It is a common belief that large meals provoke considerable postprandial reflux and it results from an increase in the rate of transient lower esophageal sphincter relaxations. One study also revealed that rapid food intake produces more gastroesophageal reflux in healthy volunteers. So this study attempted to evaluate the relationship between dietary habit and GEFV abnormality. The investigators used a questionnaire regarding the dietary habit to the population undergoing EGD in a self-paid health examination.

ELIGIBILITY:
Inclusion Criteria:

* The healthy subjects undergo EGD in a self-paid health examination in WanFang Hospital.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: healthy subjects
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Grading of Gastroesophageal Flap Valve by Esophagoduodenoscopy | 1 year
Dietary habit questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Fa Chen, M.D., Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Yung-Fa Chen, Taipei, Taipei, Taiwan